CLINICAL TRIAL: NCT04597294
Title: A Randomized, Multicenter Clinical Trial Comparing the Combination of Perioperative FLOT Chemotherapy and Preoperative Laparoscopic Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Plus Gastrectomy to Perioperative FLOT Chemotherapy and Gastrectomy Alone in Patients With Advanced Gastric Cancer at High Risk of Peritoneal Recurrence
Brief Title: Prophylactic Preoperative HIPEC in Advanced Gastric Cancer at High Risk of Peritoneal Recurrence
Acronym: CHIMERA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, MD, PhD, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Gastric CHIMERA Trial; 2020-001419-25 (EudraCT Number); 2019/ABM/01/00020-00 (Other Grant/Funding Number: Medical Research Agency)
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: HIPEC; FLOT; Gastric cancer; Lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomization 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative FLOT + prophylactic HIPEC + surgery (Experimental): After 4 doses of preoperative FLOT chemotherapy diagnostic laparoscopy will be performed - patients without distant metastases will be randomised, in those randomised to experimental arm HIPEC with irinotecan will be performed (a dose of 300 mg/m2 body surface area will be administered over 45 minutes at a temperature of 42 degrees Celsius)
  Interventions: Combination Product: FLOT + HIPEC + Surgery
- Perioperative FLOT + surgery (Active Comparator): Standard treatment regimen for advanced gastric cancer
  Interventions: Combination Product: FLOT + Surgery

INTERVENTIONS:
Combination Product: FLOT + HIPEC + Surgery — HIPEC with irinotecan after 4 doses of preoperative FLOT chemotherapy
  Other Names: Prophylactic HIPEC
  Arms: Perioperative FLOT + prophylactic HIPEC + surgery
Combination Product: FLOT + Surgery — Perioperative FLOT chemotherapy (4 doses before and 4 doses after gastrectomy) and surgery
  Other Names: Perioperative FLOT + Surgery
  Arms: Perioperative FLOT + surgery

SUMMARY:
The study was designed to evaluate the efficacy of perioperative FLOT chemotherapy in combination with perioperative hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with advanced gastric cancer at high risk of peritoneal metastases. The impact of treatment on peritoneal recurrence and survival over 6 months, 1, 3 and 5 years will be assessed.

DETAILED DESCRIPTION:
This is a randomized, multicenter, clinical trial in which 598 patients with advanced gastric cancer at high risk of peritoneal metastases are randomly allocated to receive either preoperative hyperthermic intraperitoneal chemotherapy (HIPEC) plus gastrectomy (experimental group) or gastrectomy alone (control group). All patients, regardless of allocation, will additionally receive 4 cycles of FLOT chemotherapy (docetaxel 50 mg/m2, oxaliplatin 85 mg/m2, leucovorin 200 mg/m2 and 5-fluorouracil 2600 mg/m2) before surgery ± HIPEC and 4 cycles of FLOT chemotherapy after gastrectomy. The main outcome is frequency of peritoneal recurrence by 6-months post-operative. Patients will be followed for 5 years and undergo additional evaluations at 6 months, 1 year, 3 and 5 years.

The study will take place at 7 hospitals across Poland. All participating centers have the equipment and skills to perform all necessary procedures in this study. The below centers specialize in the treatment of stomach cancer with many documented years of experience. They are trained in the maintenance of a register, possess the skills to conduct appropriate research analyses and are equipped with a system for assessing the quality of both surgical and oncological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer confirmed histopathologically in tumor specimens.
* Age 18-75 years.
* Advanced gastric cancer cT3 / cT4a / N0-3b.
* No distant metastases on computed tomography (CT) scan of the chest, abdomen and pelvis (cM0).
* Written consent to participate in the study.

Exclusion Criteria:

* No clear histopathological confirmation of gastric cancer.
* Age > 75 years.
* Poor general condition (Performance Status 3 or more on the Eastern Cooperative Oncology Group (ECOG)/World Health Organization scale).
* Previous abdominal surgery (including oncological surgery), other than laparoscopic cholecystectomy or appendectomy (open or laparoscopic).
* Pregnancy and lactation.
* Refusal to participate or an inability to provide written consent.
* Coexisting cancer in another location.
* Systemic treatment or radiotherapy for another cancer.
* Dysphagia requiring surgical treatment (gastric resection or nutritional jejunostomy) before starting neoadjuvant treatment and indication for accelerated surgery for other reasons.
* Disqualification for perioperative FLOT4 chemotherapy as decided by a multi-specialist consultation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Peritoneal recurrence rate | 6 months
  The rate of peritoneal recurrences at 6 month time from randomisation

SECONDARY OUTCOMES:
Overall survival | 6 months
  Overall survival at 6 month follow-up
Overall survival | 3 years
  Overall survival at 3 year follow-up
Overall survival | 5 years
  Overall survival at 5 year follow-up
Local recurrence rate | 3 years
  Locoregional recurrence rate at 3 year follow-up
Systemic recurrence rate | 3 years
  Systemic recurrence rate at 3 year follow-up
Local recurrence rate | 5 years
  Locoregional recurrence rate at 5 year follow-up
Systemic recurrence rate | 5 years
  Systemic recurrence rate at 5 year follow-up
Complications rate | 6 months
  According to CTCAE version 5 and Clavien-Dindo classification
Treatment-related quality of life assessed by Quality Of Life Questionnaire (QLQ) C30 version 3.0 | 6 months
  Score range 0-100, higher score represents a higher (better) level of functioning
Treatment-related quality of life assessed by Quality of Life Questionnaire-Stomach (STO22) | 6 months
  Score range 0-100, higher scores represent worse quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Richter, Professor, Study Director — Jagiellonian University
Locations (1):
- Department of General, Oncological, Gastroenterological Surgery and Transplantology, Krakow, Lesser Poland Voivodship, Poland

IPD SHARING:
Plan to Share IPD: No